CLINICAL TRIAL: NCT02057601
Title: Postoperative Analgesia Following Surgery for Fractured Neck of Femur: a Comparison of Periarticular Infiltration of Local Anaesthetic With Systemic Postoperative Analgesics
Brief Title: Postoperative Analgesia for Fractured Neck of Femur With Periarticular Infiltration of Local Anaesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Szilard Szucs, Clinical Lecturer in Anaesthesia, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECM4 (zz) 09/04/13; ECM 4 (zz) 09/04/13 (Other: Clinical Research Ethics Committee, Cork, Ireland)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Fractured Neck of Femur; Postoperative Pain
Keywords: Local anaesthetic infiltration; Fractured neck of femur; Postoperative pain
MeSH Terms: conditions — Femoral Neck Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infiltration group (Experimental): The patients in this group will receive spinal anaesthesia with intrathecal bupivacaine 0.5% 2.0ml and will receive peri-surgical site infiltration before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight with epinephrine made up to a volume of 1.5ml/kg with saline.
  Interventions: Drug: Levobupivacaine infiltration group
- Non infiltration group (No Intervention): The patients in this group will receive spinal anaesthesia with intrathecal bupivacaine 0.5% 2.0 ml.

INTERVENTIONS:
Drug: Levobupivacaine infiltration group — The patients in the intervention group will receive peri-surgical site infiltration before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight with epinephrine made up to a volume of 1.5ml/kg with saline.
  Arms: Infiltration group

SUMMARY:
The purpose of this study is to determine that periarticular levobupivacaine infiltration after surgical fixation of fractured neck of femur will improve the early postoperative pain sensation.

DETAILED DESCRIPTION:
Fractured neck of femur is a common cause of admission to hospital for elderly patients and requires operative fixation, which is usually associated with significant pain in the early postoperative period. Postoperative pain can delay mobilisation and discharge from the hospital. The administration of opioid drugs in the postoperative period is associated with significant adverse effects. Following total knee replacements local anaesthetic infiltration led to a significantly decreased duration of hospital stay due to decreased postoperative pain (1). Continuous postoperative wound infiltration after shoulder surgery with ropivacaine, (2 mg/ml and 3.75 mg/ml), results in lower pain scores and opioid requirement compared with infiltration of placebo (2). Effective pain management in the postoperative period is important to aid early mobilisation and decrease morbidity (3).

In our hospital, surgical fixation of fractured neck of femur is routinely performed under spinal anaesthesia with intrathecal bupivacaine.. This provides excellent conditions for surgery and gives satisfactory analgesia in the early postoperative period. However, clinical observation indicates that a period of inadequate analgesia often occurs after the offset of intrathecal local anaesthetic effect. Wound infiltration with local anaesthetic after total hip and knee replacement has been investigated as an alternative method of postoperative analgesia (4-8).

Hypotheses Perioperative infiltration of the surgical site with levobupivacaine (in addition to standard systemic analgesics) decreases pain during the first day after surgery.

This technique decreases post-operative systemic opioid requirements and the incidence of associated adverse effects To test these hypotheses we propose to carry out a prospective, randomized controlled clinical study in patients undergoing surgical fixation of fractured neck of femur under spinal anaesthesia.

To our knowledge, a study comparing these two techniques has not been performed previously.

Objectives To evaluate the analgesic efficacy of wound infiltration with levobupivacaine local anaesthetic with 1:200,000 epinephrine after the surgical fixation of fractured neck of femur.

Primary outcome measure Quality of analgesia at 12 hours postoperatively as assessed by verbal rating score (VRS) for pain at rest and on movement.

Methodology

Study design: A prospective, randomized clinical trial.(will be registered with Clinicaltrial.com)

Sample size: We performed a power analyis using our own previous published data, VRS (0-10) pain scores on passive movement in the 12th postoperative hour was 4.4(3.3) mean(SD). We consider that a decrease in the VAS for pain (in the intervention group of 50% would be clinically relevant. To reliably answer our question, with a power of 0.8 and a statistical significance of 0.05, we calculate that we will require a minimum of 17 patients in each group.

Patient population: Adult patients ( > 60 years) undergoing surgical fixation of fractured neck of femur.

Duration of study period: We will monitor patients perioperatively and during the postoperative period for 2 days.

Overall design: With institutional ethical approval and having obtained written informed consent, 40 patients will be randomly allocated to one of two groups using random number tables and a sealed envelope technique. The first group will receive spinal anaesthesia with intrathecal bupivacaine 0.5% 2.0 ml. The second group will receive spinal anaesthesia with intrathecal bupivacaine 0.5% 2.0ml and will receive peri-surgical site infiltration before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight with epinephrine made up to a volume of 1.5ml/kg with saline.

Both groups will be prescribed regular postoperative analgesia of paracetamol 1g qds PO/PR and diclofenac 75mg bd PO. Oxycodone ('Oxynorm') 5-10mg PO qds/prn will also be prescribed. Cyclizine 50 mg i.m. prn/tds will be prescribed for nausea and vomiting. If necessary, ondansetron 4 - 8mg i.v. prn/qds will be administered as a rescue anti-emetic.

The patients will be assessed at 2, 6, 12, 24 and 48 hours postoperatively. We will assess severity of pain using VRS at rest and on passive movement of the operative hip joint, cumulative morphine consumption, quality of analgesia during early mobilisation, compliance with physiotherapy, and adverse effects associated with opioid administration, [(i) sedation (1, awake; 2-drowsy; 3-asleep, easily rousable; 4-asleep, hard to rouse), (ii) incidence and severity of postoperative nausea (0 - no nausea, 1 - complaints of nausea but tolerable, 2 - needs cyclizine 50 mg i.m.), (iii) respiratory depression (ventilatory frequency less than 8 min-1); (iv) pruritus (1-no itch; 2-itching but tolerable; 3-severe itch needs piriton 5 mg i.m.); (v) urinary retention (C- catheterized electively postoperatively; N-no catheter required; R-catheter sited because of urinary retention)]. Patients will be asked to rate their satisfaction with perioperative pain management ( on 0-10 VRS) and whether they would have the same pain therapy again.

Statistical Analysis Collected data will be examined for normality. Quantitative data e.g. analgesic consumption and visual analog pain scores will be examined using the Student-t test. Categorical data will be examined using the chi-squared test. Fisher's Exact test will be used to compare non-parametric data (i.e. necessity of a urinary catheter). P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgical fixation of fractured neck of femur
* consent to spinal anaesthesia
* ASA grade 1-3

Exclusion Criteria:

* Patients refusal
* Mini mental scores less than 25
* Allergy to bupivacaine, morphine, paracetamol and diclofenac
* Skin lessons/ infections at the site of injection
* Uncorrected renal dysfunction
* Coagulation disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
VRS pain score on passive movement 12 hours after the surgery | 12 hours after the surgery
  We will assess the patients 12 hours after the surgical fixation of fractured neck of femur on passive movement (elevating the limb with 30 degree)

SECONDARY OUTCOMES:
VRS pain scores in the first two postoperative day. | 48 hours
  After the operative fixation of fractured neck of femur, the patients will be assessed in the second, sixth, 12th, 24th and 48th postoperative hour. We will using VRS (0-10) pain scores at rest and passive movement.

OTHER OUTCOMES:
Haemodynamic parameters | 48 hour
  After surgical fixation of fractured neck of femur, the patients will be assessed in the second, sixth, 1 2nd, 24th and 48th hour. Blood pressure, heart rate, reap rate will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland